CLINICAL TRIAL: NCT04967508
Title: A Phase III, Randomised, Double-blind, Multicentre Clinical Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Immunogenicity of SB17 (Proposed Ustekinumab Biosimilar) Compared to Stelara® in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Compare SB17 (Proposed Ustekinumab Biosimilar) to Stelara® in Subject With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB17-3001
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Psoriasis; Moderate to Severe Plaque Psoriasis
Keywords: Psoriasis; Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SB17 (Proposed Ustekinumab Biosimilar) (Experimental)
  Interventions: Drug: SB17 (Proposed Ustekinumab Biosimilar)
- Stelara® (Ustekinumab) (Active Comparator)
  Interventions: Drug: Stelara® (Ustekinumab); Drug: SB17 (Proposed Ustekinumab Biosimilar)

INTERVENTIONS:
Drug: Stelara® (Ustekinumab) — Subjects randomised into Stelara® group will receive Stelara® (45 mg) via subcutaneous injection at Week 0, 4, and then every 12 weeks up to Week 40.
  Arms: Stelara® (Ustekinumab)
Drug: SB17 (Proposed Ustekinumab Biosimilar) — Subjects randomised into SB17 group will receive SB17 (45 mg) via subcutaneous injection at Week 0, 4, and then every 12 weeks up to Week 40.
  Starting at Week 28, subjects transited from Stelara® to SB17 will receive SB17 via subcutaneous injection.

SUMMARY:
This is a randomised, double-blind, multicentre clinical study to evaluate the efficacy, safety, tolerability, PK, and immunogenicity of SB17 compared to Stelara® in subjects with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
Subjects will be randomised in a 1:1 ratio to receive either SB17 or Stelara® via subcutaneous injection. At Week 28, subjects receiving Stelara® will be randomised again in a 1:1 ratio to either continue on Stelara® or be transitioned to SB17. Investigational products (IPs) (SB17 or Stelara®) will be administered at Week 0, 4, and then every 12 weeks up to Week 40, and the last assessment will be done at Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older at Screening.
* Have plaque psoriasis diagnosed at least 6 months, with or without psoriatic arthritis.
* Have plaque psoriasis with the involvement and severity of total affected BSA ≥ 10%, PASI score of ≥ 12 and PGA score of ≥ 3 (moderate).
* Considered to be a candidate for phototherapy or systemic therapy for psoriasis
* Less than 95 kg of body weight.
* Adequate hematological, renal and hepatic function by central lab.
* Non-childbearing potential female, or childbearing potential female subjects or male subjects with their partners who agree to use at least two forms of appropriate contraception method from Screening until 15 weeks after the last dose of IP.

Exclusion Criteria:

* Have nonplaque forms of psoriasis, including erythrodermic, pustular, guttate, or drug-induced psoriasis.
* Have other skin disease than psoriasis that requires topical or systemic corticosteroids.
* Prior biologic use as any TNF inhibitors within the previous 6 months; any IL-12 or IL-23 inhibitor biologics, IL-17 inhibitor, rituximab, or integrin inhibitor biologics at any time; or other biologics within the longer of either 5 half-lives or 3 months prior to randomisation.
* Known allergic reactions or hypersensitivity to ustekinumab or to any ingredients of Stelara® or SB17
* History of exfoliative dermatitis, reversible posterior leukoencephalopathy syndrome, facial palsy, allergic alveolitis, or non-infectious pneumonia.
* Have received phototherapy or conventional systemic therapy for psoriasis within 4 weeks prior to Randomisation.
* Have received topical therapy for psoriasis within 2 weeks prior to Randomisation.
* Women who are pregnant or nursing at Screening, or men and women planning pregnancy during the study period and until 15 weeks after the last dose of IP.
* Have received a live or live attenuated viral vaccine or a live bacterial vaccine within 4 weeks (for BCG, 12 months) prior to Randomisation.
* Have active or latent tuberculosis.
* History of ongoing infection or a positive test of HBV, HCV, or HIV infection
* History of sepsis, chronic or recurrent infection
* History of malignancy within the last 5 years
* History of lymphoproliferative disease or leukemia
* History of myocardial infarction, NYHA III/IV congestive heart failure, or stroke within 12 months
* Have uncontrolled hypertension or diabetes
* History of uncontrolled psychiatric disorders or risk of suicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-11-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- Czechia (4):
  - SB Investigative Site, Brno
  - SB Investigative Site, Ostrava
  - SB Investigative Site, Pardubice
  - SB Investigative Site, Prague
- Estonia (2):
  - SB investigative site, Tallinn
  - SB Investigative Site, Tartu
- SB Investigative Site, Zalaegerszeg, Hungary
- Latvia (2):
  - SB Investigative Site, Riga
  - SB Investigative Site, Talsi
- Lithuania (2):
  - SB Investigative Site, Kaunas
  - SB Investigative Site, Vilnius
- Poland (10):
  - SB Investigative Site, Elblag
  - SB Investigative Site, Kielce
  - SB Investigative Site, Krakow
  - SB Investigative Site, Lodz
  - SB Investigative Site, Lublin
  - SB Investigative Site, Rzeszów
  - SB Investigative Site, Siedlce
  - SB Investigative Site, Skierniewice
  - SB Investigative Site, Świdnik
  - SB Investigative Site, Warsaw
- South Korea (2):
  - SB Investigative Site, Seongnam
  - SB Investigative Site, Suwon
- Ukraine (9):
  - SB Investigative Site, Dnipro
  - SB Investigative Site, Kharkiv
  - SB Investigative Site, Kherson
  - SB Investigative Site, Kyiv
  - SB Investigative Site, Lviv
  - SB Investigative Site, Odesa
  - SB Investigative Site, Uzhhorod
  - SB Investigative Site, Vinnytsia
  - SB Investigative Site, Zaporizhzhia

RESULTS

PARTICIPANT FLOW:
Groups:
- SB17 (Proposed Ustekinumab Biosimilar): Subjects were randomised into SB17 (Proposed Ustekinumab Biosimilar) group to receive SB17 (45 mg) via subcutaneous injection at Week 0, 4, and then every 12 weeks until Week 28 (i.e., Week 0, Week 4, and Week 16).
  At Week 28, subjects in the SB17 group were re-randomised (to maintain blindness) but continued to receive SB17 during the transition period (i.e., Week 28 and Week 40).
- Stelara (Ustekinumab): Subjects were randomised into Stelara (Ustekinumab) group to receive Stelara (45 mg) via subcutaneous injection at Week 0, 4, and then every 12 weeks until Week 28 (i.e., Week 0, Week 4, and Week 16).
  At Week 28, subjects in the Stelara (Ustekinumab) group were re-randomised and either transitioned to SB17 or continued to receive Stelara during the transition period (i.e., Week 28 and Week 40).
- Stelara to SB17: Subjects, who were randomised at Week 0 to receive Stelara (Ustekinumab) in the Main Period, were re-randomised at Week 28 to receive SB17 once every 12 weeks during the transition period (i.e., Week 28 and Week 40).
- Stelara to Stelara: Subjects, who were randomised at Week 0 to receive Stelara (Ustekinumab) in the Main Period, were re-randomised at Week 28 to receive Stelara (Ustekinumab) once every 12 weeks during the transition period (i.e., Week 28 and Week 40).
Period: Main Period
Arm/Group | SB17 (Proposed Ustekinumab Biosimilar) | Stelara (Ustekinumab) | Stelara to SB17 | Stelara to Stelara
Started | 249 | 254 | 0 | 0
Completed | 237 | 244 | 0 | 0
Not Completed | 12 | 10 | 0 | 0
Period: Transition Period
Arm/Group | SB17 (Proposed Ustekinumab Biosimilar) | Stelara (Ustekinumab) | Stelara to SB17 | Stelara to Stelara
Started | 237 | 0 | 122 (Subjects, who were randomised at Week 0 to receive Stelara (Ustekinumab) in the Main Period, were re-randomised at Week 28 to receive SB17 once every 12 weeks during the transition period (i.e., Week 28 and Week 40)) | 122 (Subjects, who were randomised at Week 0 to receive Stelara (Ustekinumab) in the Main Period, were re-randomised at Week 28 to receive Stelara (Ustekinumab) once every 12 weeks during the transition period (i.e., Week 28 and Week 40).)
Completed | 233 | 0 | 117 | 116
Not Completed | 4 | 0 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB17 (Proposed Ustekinumab Biosimilar) | Stelara (Ustekinumab) | Total
Number analyzed (Participants) | 249 | 254 | 503
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 234 | 234 | 468
  >=65 years | 15 | 19 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (13.21) | 44.3 (12.42) | 44.2 (12.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 92 | 191
  Male | 150 | 162 | 312
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Korean | 2 | 4 | 6
  Ethnicity: Mixed Ethnicity | 0 | 1 | 1
  Ethnicity: Other | 247 | 249 | 496
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2 | 4 | 6
  Race: White | 247 | 250 | 497
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 27.2 (3.94) | 26.8 (3.66) | 27.0 (3.81)
Total psoriasis BSA involvement [Mean (Standard Deviation); unit: %] | 27.3 (13.49) | 26.7 (13.77) | 27.0 (13.62)
Duration of psoriasis [Mean (Standard Deviation); unit: years] | 15.0 (11.38) | 16.1 (11.88) | 15.6 (11.64)
PASI at baseline [Mean (Standard Deviation); unit: index] | 22.5 (7.82) | 22.1 (7.69) | 22.3 (7.75)
PGA Score of ≥ 4 (Marked or Severe) at baseline [Count of Participants; unit: Participants] | 92 | 94 | 186
Dermatology Life Quality Index (DLQI) at baseline [Mean (Standard Deviation); unit: scores on a scale] — DLQI score ranges from 0 to 30 (a lower score means better quality of life).
  scores on a scale | 13.4 (7.24) | 13.2 (6.96) | 13.3 (7.09)
History of psoriatic arthritis [Count of Participants; unit: Participants]
  Yes | 64 | 54 | 118
  No | 185 | 200 | 385

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in PASI at Week 12
Description: Psoriasis area severity index (PASI) measures the activity of psoriasis through erythema, induration and scaling and can range from 0 to 72. The degree of PASI improvement in terms of percent change from baseline at Week 12 is measured.
Time Frame: Baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | SB17 (Proposed Ustekinumab Biosimilar) | Stelara (Ustekinumab)
Number analyzed (Participants) | 243 | 249
Percent change | 85.7 (2.53) | 86.3 (2.41)

ADVERSE EVENTS:
Time Frame: Overall Period (up to 52 weeks)
Arm/Group | SB17 (Proposed Ustekinumab Biosimilar) | Stelara (Ustekinumab) | Stelara to SB17 | Stelara to Stelara
All-Cause Mortality (participants affected / at risk) | 0/249 | 0/254 | 0/122 | 0/122
Serious Adverse Events (participants affected / at risk) | 7/249 | 6/254 | 2/122 | 3/122
Other Adverse Events (participants affected / at risk) | 50/249 | 62/254 | 28/122 | 31/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB17 (Proposed Ustekinumab Biosimilar) (N=249) | Stelara (Ustekinumab) (N=254) | Stelara to SB17 (N=122) | Stelara to Stelara (N=122)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pelvic adhesions (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB17 (Proposed Ustekinumab Biosimilar) (N=249) | Stelara (Ustekinumab) (N=254) | Stelara to SB17 (N=122) | Stelara to Stelara (N=122)
Nasopharyngitis (Infections and infestations) | 23 (26) | 23 (30) | 12 (16) | 10 (12)
COVID-19 (Infections and infestations) | 18 (19) | 29 (29) | 12 (12) | 15 (15)
Upper respiratory tract infection (Infections and infestations) | 12 (15) | 16 (19) | 8 (10) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT04967508/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT04967508/SAP_001.pdf